CLINICAL TRIAL: NCT01796106
Title: Clinical Efficacy of Caries Infiltration (Icon) - A Randomized, Blinded and Controlled Pilot Study of Early Caries Progression Detection
Brief Title: Clinical Trial Proximal Caries Infiltration and Detection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment slower than expected.
Sponsor: DMG Dental Material Gesellschaft mbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DETECT13
Record Dates: First submitted 2012-11-01; First posted 2013-02-21 (Estimated); Results first posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-06

CONDITIONS: Caries,Dental
Keywords: Caries infiltration; Resin infiltration; Caries progression; Icon
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resin infiltration (Experimental): Enrolled proximal early caries lesions will be treated using the resin infiltrant Icon (DMG, Germany).
  Interventions: Device: Resin infiltration
- Fluoride varnish & Oral hygiene instruction (Active Comparator): Oral hygiene instruction and topical fluoridation therapy (Duraphat Fluoride Varnish, Colgate, USA) will be provided.
  Interventions: Device: Fluoride varnish & Oral hygiene instruction

INTERVENTIONS:
Device: Resin infiltration — Up to two proximal early caries lesions (only if the second lesion is in a separate quadrant) per participant will be included. After radiographic and SFE imaging to assess lesion depth, the study lesions will be treated using the resin infiltrant Icon (DMG, Germany) according to manufactures´ instructions. Essentially, the treatment consists of the following parts: 1) isolating the tooth with a rubber dam and cleaning its surface; 2) removing/ conditioning the surface layer of the lesion (using Icon-Etch) to open the lesion body; 3) drying of the exposed porous enamel; 4) infiltrating the existing pore volume with the resin infiltrant (Icon Infiltrant); 5) light curing of the resin infiltrant; 6) repeating the infiltration step including light curing; followed by 7) finalizing using interproximal finishing/polishing strips.
  Other Names: Icon (DMG, Germany), approximal resin infiltration kit
  Arms: Resin infiltration
Device: Fluoride varnish & Oral hygiene instruction — Up to two proximal early caries lesions (only if the second lesion is in a separate quadrant) per participant will be included. After radiographic and SFE imaging to assess lesion depth oral hygiene instruction and topical fluoridation therapy will be provided. For topical fluoridation Duraphat Fluoride Varnish (Colgate, USA) will be used according to manufactures´ instructions.
  Other Names: Duraphat Fluoride Varnish (Colgate, USA)
  Arms: Fluoride varnish & Oral hygiene instruction

SUMMARY:
The purpose of this study is to investigate the clinical efficacy of resin infiltration (Icon, DMG, Germany) compared to fluoride varnish (Duraphat Fluoride Varnish, Colgate, USA) in the management of proximal early caries lesions in primary molars over 24 months. In addition, this study will assess the use of a scanning fiber endoscope (SFE) laser optical device for the assessment of caries lesions and their progression in comparison to radiographic examination.

A total of 50 participants (age 6-13 years) with at least 1 proximal early caries lesion will be enrolled. The participants will be followed up at 12 and 24 months. Lesion status will be monitored through radiographic and SFE laser optical device imaging.

DETAILED DESCRIPTION:
Introduction: Dental caries remains one of the most prevalent diseases worldwide. It is a dynamic process that causes destruction of tooth structure by dissolving the enamel. While it is possible to restore the structure and function of the tooth by placing a filling, it is preferable to slow down or reverse the caries process at an early state. Proximal surfaces are hereby particularly susceptible to caries as the contact area between teeth is difficult to access. While non-invasive techniques such as remineralization (using topical fluoride) or biofilm control are options to manage early caries lesions, their effectiveness may be compromised due to poor patient compliance. Alternatives are micro-invasive strategies such as resin infiltration, whereby a highly viscous resin is infiltrated into the porous enamel of caries lesions to erect an internal barrier that blocks acid diffusion, thereby inhibiting caries lesion progression.

Another important aspect in caries management is diagnostic, with visual-tactile examination and radiographs being standard of care. However, visual-tactile techniques are known to be unreliable due to subjectivity and fail to differentiate between varies stages of caries progression. Caries diagnostic is thus assisted by radiographic imaging, which however, also has a limited sensitivity and requires the use of x-rays. While alternatives for caries imaging have been developed (e.g. quantitative laser or light fluorescence (QLF) or electrical conductance measurements (ECM)) no gold standard could be established so far highlighting the need for new save and sensitive imaging techniques.

Objective: To assess the clinical efficacy of resin infiltration (Icon, DMG, Germany) compared to fluoride varnish (Duraphat Fluoride Varnish, Colgate, USA) in the management of proximal early caries lesions over 24 months. In addition, the use of a SFE laser optical device for the assessment of caries lesions and their progression will be assessed in comparison to radiographic examination.

Materials and Methods: 50 volunteers (age 6-13 years) with at least 1 proximal early caries lesion in primary molars will be enrolled and randomly assigned to the resin infiltration and control groups. In the resin infiltration group early caries lesions will be treated using Icon (DMG), whereas the lesions in the control group will be managed using Oral Hygiene Instructions (OHI) and topical fluoridation (Duraphat Fluoride Varnish, Colgate). Lesion depth will be assessed through radiographic evaluation as well as through a novel optical device based on scanning fiber endoscope (SFE) technology for early caries detection through laser light imaging. SFE laser optical device prototypes developed by the University of Washington's Human Photonics Lab (HPL) will be utilized. Such a device is already in human use for applications such as imaging and cancer screening.

Clinical Significance: Resin infiltration of early caries lesions may be an effective therapeutic strategy in paediatric dentistry to reduce caries progression. Additionally, the SFE optical device may be suitable technology to visualize early caries lesions and their progression, which would offer a safe alternative to radiography for assessing and monitoring dental caries.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-13 years
* Early caries lesions in primary molars (depth: E1 or E2)
* Good general health
* Available for 12 & 24 months recalls
* Signed consent/assent/HIPAA

Criteria used to assess teeth for acceptance into this study:

* Teeth fully erupted, in functional occlusion and
* Radiographic evidence of early caries in interproximal areas

Exclusion Criteria:

* Participation in other study
* History of adverse reaction on clinical material
* Sensitivity during screening test
* Poor access to teeth
* Patient refusing radiographic examination

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Berg, DDS, MS, Principal Investigator — The Center for Pediatric Dentistry
Locations (1):
- The Center for Pediatric Dentistry, Seattle, Washington, United States

REFERENCES:
- [Background] Anusavice KJ. Present and future approaches for the control of caries. J Dent Educ. 2005 May;69(5):538-54. PMID 15897335

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from patients seeking treatment at the Center for Pediatric Dentistry Seattle, Washington, USA. The first participant was enrolled in March 2015 and the last was enrolled in March 2016.
Pre-assignment Details: Up to two proximal early caries lesions per participant were included, but only if the second lesion was located in a separate quadrant.
Units Other Than Participants: Lesions
Groups:
- Resin Infiltration: After radiographic and scanning fiber endoscope (SFE) imaging to assess lesion depth, the study lesions were treated using the resin infiltrant Icon (DMG, Germany) according to manufactures´ instructions.
- Fluoride Varnish & Oral Hygiene Instruction: After radiographic and scanning fiber endoscope (SFE) imaging to assess lesion depth oral hygiene instruction and topical fluoridation therapy were provided. For topical fluoridation Duraphat Fluoride Varnish (Colgate, USA) has been used according to manufactures´ instructions.
Period: Overall Study
Arm/Group | Resin Infiltration | Fluoride Varnish & Oral Hygiene Instruction
Started | 5; 5 Lesions | 7; 7 Lesions
12 Months Follow up | 0; 0 Lesions | 0; 0 Lesions
Completed (24 month follow up was expected for completion.) | 0; 0 Lesions | 0; 0 Lesions
Not Completed | 5; 5 Lesions | 7; 7 Lesions
Not completed — Study was terminated due to insufficient recruitment before follow ups could be completed | 5 | 7

BASELINE CHARACTERISTICS:
Units Other Than Participants: Lesions
Groups:
- Resin Infiltration: After radiographic and SFE imaging to assess lesion depth, the study lesions were treated using the resin infiltrant Icon (DMG, Germany) according to manufactures´ instructions.
- Fluoride Varnish & Oral Hygiene Instruction: After radiographic and SFE imaging to assess lesion depth oral hygiene instruction and topical fluoridation therapy were provided. For topical fluoridation Duraphat Fluoride Varnish (Colgate, USA) has been used according to manufactures´ instructions.
- Total: Total of all reporting groups
Arm/Group | Resin Infiltration | Fluoride Varnish & Oral Hygiene Instruction | Total
Number analyzed (Participants) | 5 | 7 | 12
Number analyzed (Lesions) | 5 | 7 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 7 | 12
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 0 | 0 | 0
  Unknown | 5 | 7 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Caucasian | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0
  Other | 0 | 0 | 0
  Unknown | 5 | 7 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 7 | 12
Lesion size [Count of Units; unit: Lesions] — Categorical lesion depth as measured by radiographs. E1 (lesion within the outer half of enamel), E2 (inner half of enamel), D1 (outer third of dentin), D2 (middle third of dentin).
  Lesions
    E1 | 2 | 3 | 5
    E2 | 2 | 4 | 6
    D1 | 1 | 0 | 1
    D2 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Lesions That Changed in Size (E1->E2->D1->D2-> Filling)
Description: Change in categorical lesion depth (progression to next depth category lesion; E1->E2->D1->D2->filling) as measured by pairwise comparison of radiographs (baseline versus follow up time point). E1 (lesion within the outer half of enamel), E2 (inner half of enamel), D1 (outer third of dentin), D2 (middle third of dentin).
Time Frame: 24 months
Population: This study was terminated due to insufficient recruitment. The 24 month follow up was not reached for any enrolled participant at the time of termination.
Units Other Than Participants: Lesions
Arm/Group | Resin Infiltration | Fluoride Varnish & Oral Hygiene Instruction
Number analyzed (Participants) | 0 | 0
Number analyzed (Lesions) | 0 | 0

2. Secondary Outcome: Validation of SFE Imaging for Lesion Size Assessment: SFE Imaging vs. Radiographic Imaging
Description: Categorical lesion depth (E1, E2, D1, D2) is measured using SFE imaging. The results are compared to the assessment of categorical lesion depth using radiographic imaging (state of the art method). Outcomes are defined as follows: 1) positive (if SFE imaging gave the same result as the radiograph analysis), 2) negative (if SFE imaging gave a different result as the radiograph analysis) and 3) failure (if lesion depth could not be assessed using SFE imaging).
  Categorical lesion depth: E1 (lesion within the outer half of enamel), E2 (inner half of enamel), D1 (outer third of dentin), D2 (middle third of dentin).
Time Frame: 0, 12 and 24 months
Population: This study was terminated due to insufficient recruitment. Only 12 (out 50 planned) participants could be recruited and the 12 and 24 month follow ups were not reached for any enrolled participant at the time of termination.
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Resin Infiltration | Fluoride Varnish & Oral Hygiene Instruction
Number analyzed (Participants) | 5 | 7
Number analyzed (Lesions) | 5 | 7
Lesions
  Baseline: Positive | 1 | 2
  Baseline: Negative | 1 | 2
  Baseline: Failure | 3 | 3
  12 months: number analyzed (Participants) | 0 | 0
  12 months: number analyzed (Lesions) | 0 | 0
  12 months: Positive | 0 | 0
  12 months: Negative | 0 | 0
  12 months: Failure | 0 | 0
  24 months: number analyzed (Participants) | 0 | 0
  24 months: number analyzed (Lesions) | 0 | 0
  24 months: Positive | 0 | 0
  24 months: Negative | 0 | 0
  24 months: Failure | 0 | 0

3. Secondary Outcome: Number of Lesions That Changed in Size (E1->E2->D1->D2-> Filling)
Description: as for outcome 1
Time Frame: 12 months
Population: This study was terminated due to insufficient recruitment. The 12 month follow up was not reached for any enrolled participant at the time of termination.
Units Other Than Participants: Lesions
Arm/Group | Resin Infiltration | Fluoride Varnish & Oral Hygiene Instruction
Number analyzed (Participants) | 0 | 0
Number analyzed (Lesions) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 12 months. Data were collected for each participant from inclusion until this study was terminated (just before the 12 month follow up was reached for the first participant). Consequently, the specific time period varies for each participant depending on the time of inclusion as follows: Group 1: Resin Infiltration: 12, 10, 6, 4 and 2 months Group 2: Fluoride Varnish & Oral Hygiene Instruction: 11, 9, 9, 5, 4, 1 and <1 month
Arm/Group | Resin Infiltration | Fluoride Varnish & Oral Hygiene Instruction
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/7
Other Adverse Events (participants affected / at risk) | 0/5 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-13): https://cdn.clinicaltrials.gov/large-docs/06/NCT01796106/Prot_SAP_000.pdf